CLINICAL TRIAL: NCT03923426
Title: REAL-WORLD OBSERVATIONAL STUDY OF ZAVICEFTA (REGISTERED) (CEFTAZIDIME-AVIBACTAM) TO CHARACTERIZE USE PATTERNS, EFFECTIVENESS AND SAFETY - EZTEAM STUDY
Brief Title: Real-World Observational Study Of Zavicefta to Characterize Use Patterns
Acronym: EZTEAM
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3591031; EZTEAM STUDY (Other: Alias Study Number)
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-01

CONDITIONS: Infection
Keywords: ceftazidime-avibactam; Zavicefta
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Other: Zavicefta Treatment — Non-interventional - Retrospective Chart Review

SUMMARY:
This is a non-interventional medical chart review study aiming to examine the treatment patterns, effectiveness, and safety of ceftazidime-avibactam in approximately 12 countries (including but not limited to Austria, France, Germany, Greece, Italy, Spain, United Kingdom, Russia, Argentina, Colombia, Brazil, and Mexico), with possible expansion to other countries as ceftazidime-avibactam is launched. Eligible patients are adults who have been treated with ceftazidime-avibactam in routine practice at participating sites since 01 January, 2018 onwards or since the date of launch in the country if it is posterior to 01 January, 2018. As this is an observational study, patients will be treated based on the standard of care at the discretion of their physician. No drugs will be supplied for this study and patients will receive treatment through standard local practice.

DETAILED DESCRIPTION:
This observational study will include approximately 700 hospitalized patients with a gram-negative infection, who have received at least one dose of ceftazidime-avibactam.

Patients will be recruited in approximately 62 sites across 12 countries in Europe (including Russia) and Latin America. Patients will be followed from ceftazidime-avibactam initiation until 60 days post hospital discharge, mortality, withdrawal from the study, or loss-to-follow-up, whichever occurs first.

Data will be abstracted from medical records using an electronic case report form (eCRF). Baseline data include patient socio-demographics, medical history, and clinical and microbiological characteristics of the infection treated.

Follow-up data will include details of treatment over time and clinical, microbiological, and healthcare resource utilization outcomes.

Evaluation of clinical success will be performed in patients with at least ≥72 hours of exposure to ceftazidime-avibactam.

Safety will be evaluated in all patients exposed to at least one dose of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patient ≥18 years old or considered an adult in accordance with the age of majority in the participant's country of residence at the time of treatment with ceftazidime-avibactam.
2. Patient received ≥1 dose of ceftazidime-avibactam in routine practice at participating site since 01 January, 2018 onwards or since the date of launch in the country if it is after 01 January, 2018.
3. Patient underwent microbiologic sampling ≤5 days before the initiation of ceftazidime-avibactam (irrespective of results and actual bacteriological identification).
4. Patient has all required essential data elements which include:

   1. Start and stop dates of ceftazidime-avibactam,
   2. Start and stop dates of prior antibiotic therapy used for the index infection,
   3. Type of combined antibiotic therapy (if applicable) and start and stop dates of any antibiotic combined with ceftazidime-avibactam.
5. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study where required by local regulations.

Exclusion Criteria:

Patients must not meet any of the following exclusion criteria to be eligible:

1. The patient is enrolled in any clinical trial of an investigational product. Patients who are enrolled in non-interventional studies (NISs) (e.g. registries) are eligible for inclusion.
2. The patient has received ceftazidime-avibactam in a compassionate care program setting.
3. The patient was exposed to ceftazidime-avibactam before use for the index infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with ≥72 hours of exposure to ceftazidime-avibactam at 42 European sites. Patients will be identified over a 12-month period and information about treatment will be abstracted from medical records after treatment completion. Patients will be followed from ceftazidime-avibactam initiation until 60 days post hospital discharge, mortality, withdrawal, or loss-to-follow-up, whichever occurs first.
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- Argentina (6):
  - Hospital Aleman, Buenos Aires
  - Hospital Britanico de Buenos Aires, CABA
  - CEMIC, Ciudad Autonoma Buenos Aires
  - Hospital Italiano, Ciudad Autonoma Buenos Aires
  - Hospital Privado Centro Medico de Cordoba S.A., Córdoba
  - Sanatorio Britanico S.A., Rosario
- AKH - Medizinische Universität Wien, Vienna, Austria
- Brazil (5):
  - Hospital Felício Rocho, Belo Horizonte
  - Hospital Vera Cruz, Belo Horizonte
  - CEPETI - Centro de Estudos e Pesquisa em Emergências Médicas e Terapia Intensiva, Curitiba
  - Hospital Moinho de Ventos, Porto Alegre
  - Hospital de Caridade de Santa Maria -HCAA, Santa Maria
- Colombia (4):
  - Centro médico Imbanaco, Cali
  - Caja de Compensacion Familiar de Caldas / Confa, Manizales
  - Promotora Medica Las Americas SA, Medellín
  - IPS Universitaria, Medellín
- France (5):
  - CHU Angers - Hôpital Hôtel Dieu, Angers
  - CHU Nantes - Hôtel Dieu pt, Nantes
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Centre Hospitalier de Tourcoing, Tourcoing
- Germany (2):
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - University Hospital Jena, Jena
- Greece (2):
  - University of Patras Medical School, Pátrai, Achaia
  - General Hospital of Athens Laiko, Athens, Attica
- Italy (5):
  - Policlinico Universitario Agostino Gemelli, Rome, ROMA
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria San Martino, Genoa
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Ospedale Amedeo di Savoia, Torino
- Russia (6):
  - Regional Clinical Hospital #1, Krasnodar
  - SBIH of Moscow City Clinical Hospital # 7, Moscow
  - FSBI "State Scientific Centre of Coloproctology" of the MoH of RF, Moscow
  - FSBI "Hematological Research Center" MoH of RF, Moscow
  - North-West Federal Medical Research Center n.a. V.A. Almazov, Saint Petersburg
  - SBIH Republican Clinical Hospital n.a. G. G. Kuvatov, Ufa
- Spain (5):
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hopsital Ramón y Cajal, Madrid
- United Kingdom (4):
  - Manchester University NHS Foundation Trust, Manchester, Greater Manchester
  - Sheffield Teaching Hospitals, Sheffield, South Yorkshire
  - Kings College Hospital NHS Foundation Trust, London
  - Chelsea and Westminster Hospital, London

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Soriano A, Montravers P, Bassetti M, Klyasova G, Daikos G, Irani P, Stone G, Chambers R, Peeters P, Shah M, Hulin C, Albuquerque N, Basin E, Gaborit B, Kourbeti I, Menichetti F, Perez-Rodriguez MT, Pletz MW, Sanchez M, Trompa I, Verma A, de Figueiredo MLN, Charbonneau C. The Use and Effectiveness of Ceftazidime-Avibactam in Real-World Clinical Practice: EZTEAM Study. Infect Dis Ther. 2023 Mar;12(3):891-917. doi: 10.1007/s40121-023-00762-9. Epub 2023 Feb 10. PMID 36763243
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3591031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were hospitalized with gram-negative infection and received at least one dose of ceftazidime-avibactam in routine clinical practice since 01-Jan-2018 were included in this chart review study. Participants were recruited across Europe and Latin America and were followed from ceftazidime-avibactam initiation until 60 days post hospital discharge, mortality, withdrawal from the study, or loss-to-follow-up, whichever occurred first.
Pre-assignment Details: Data was abstracted from medical records and evaluated over approximately 40 months of this study.
Groups:
- Ceftazidime-avibactam: Eligible participants who were hospitalized with gram negative infections and received at least one dose of ceftazidime-avibactam in routine clinical practice since 01-Jan-2018 were included in this chart review study.
Period: Overall Study
Arm/Group | Ceftazidime-avibactam
Started (All enrolled) | 572
Full Analysis Set (All eligible participants among enrolled) | 569
Completed (Followed through medical records up to 60 days after hospital discharge) | 417
Not Completed | 155
Not completed — Other | 19
Not completed — Lost to Follow-up | 16
Not completed — Death | 107
Not completed — Incomplete response to question | 13

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all those enrolled participants who met the study eligibility criteria. Baseline characteristics were analyzed and reported for FAS72+ which included FAS participants with at least 72 hours of exposure to ceftazidime-avibactam and FAS72- which included FAS participants with less than (<) 72 hours of exposure to ceftazidime-avibactam.
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 569
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Years
    FAS72+: number analyzed (Participants) | 516
    FAS72+ | 58.3 (18.37)
    FAS72-: number analyzed (Participants) | 53
    FAS72- | 59.7 (17.99)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Participants
    FAS72+: number analyzed (Participants) | 516
    FAS72+: Female | 164
    FAS72+: Male | 352
    FAS72-: number analyzed (Participants) | 53
    FAS72-: Female | 20
    FAS72-: Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and ethnicity were not collected Population: Race and Ethnicity were not collected from any participant.
Number of Participants According to Their Employment Status [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set.
  Participants
    number analyzed (Participants) | 516
    Full Time | 78
    Part Time | 5
    Unemployed | 67
    Retired | 159
    Not Available | 207
Height: FAS72+ Analysis set [Mean (Standard Deviation); unit: Centimeter (cm)] — Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the baseline characteristic.
  Centimeter (cm)
    number analyzed (Participants) | 358
    (all) | 169.9 (9.35)
Weight: FAS72+ Analysis set [Mean (Standard Deviation); unit: Kilogram (kg)] — Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the baseline characteristic.
  Kilogram (kg)
    number analyzed (Participants) | 368
    (all) | 76.0 (19.15)
Number of Participants With Prior Hospitalizations Within 90 days Prior to Current Hospitalization [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the baseline characteristic.
  Participants
    number analyzed (Participants) | 511
    (all) | 253
Number of Participants With Antibiotic Exposure Within 90 Days Prior to Index Hospitalization [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the baseline characteristic.
  Participants
    number analyzed (Participants) | 511
    (all) | 260
Number of Participants With any Healthcare Procedure Within 30 Days Prior to Index Date [Count of Participants; unit: Participants] — Index date was defined as start date of ceftazidime-avibactam. Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the baseline characteristic.
  Participants
    number analyzed (Participants) | 512
    (all) | 311
Number of Participants According to Antibiotic Class Used Prior to Ceftazidime-Avibactam Initiation [Count of Participants; unit: Participants] — One participant could have received more than one antibiotic. Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the baseline characteristic.
  Participants
    Aminoglycosides: number analyzed (Participants) | 259
    Aminoglycosides | 49
    Carbapenems: number analyzed (Participants) | 259
    Carbapenems | 118
    Cephalosporins: number analyzed (Participants) | 259
    Cephalosporins | 73
    Fluoroquinolones: number analyzed (Participants) | 259
    Fluoroquinolones | 65
    Glycopeptides: number analyzed (Participants) | 259
    Glycopeptides | 81
    Glycylcycline: number analyzed (Participants) | 259
    Glycylcycline | 17
    Lipopeptides: number analyzed (Participants) | 259
    Lipopeptides | 17
    Macrolides: number analyzed (Participants) | 259
    Macrolides | 24
    Monobactam: number analyzed (Participants) | 259
    Monobactam | 5
    Nitroimidazole: number analyzed (Participants) | 259
    Nitroimidazole | 26
    Other agents: number analyzed (Participants) | 259
    Other agents | 65
    Oxazolidinones: number analyzed (Participants) | 259
    Oxazolidinones | 27
    Penicillins: number analyzed (Participants) | 259
    Penicillins | 18
    Penicillins and beta-lactamase inhibitors: number analyzed (Participants) | 259
    Penicillins and beta-lactamase inhibitors | 110
    Tetracycline: number analyzed (Participants) | 259
    Tetracycline | 9
    Uncoded: number analyzed (Participants) | 259
    Uncoded | 48
Number of Participants According to Country Travelled Within the Past 3 Months [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for this baseline characteristic who travelled to other countries.
  Participants
    number analyzed (Participants) | 8
    Egypt | 1
    Germany | 1
    Italy | 1
    Netherlands | 1
    Pakistan | 1
    Spain | 2
    Turkey | 1
Number of Participants With Reported Pregnancy [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set.
  Participants
    number analyzed (Participants) | 516
    (all) | 3
Number of Weeks of Gestation Since Last Menstrual Period [Mean (Standard Deviation); unit: Weeks] — In this baseline characteristic number of weeks of gestation since last menstrual period is reported in mean. Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Weeks
    number analyzed (Participants) | 3
    (all) | 29.7 (8.39)
Number of Participants With Alcohol use [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set.
  Participants
    number analyzed (Participants) | 516
    (all) | 41
Number of Alcoholic Drinks per Week: FAS72+ Analysis set [Mean (Standard Deviation); unit: Drinks per week] — In this baseline characteristic number of alcoholic drinks per week is reported in mean. Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the baseline characteristic.
  Drinks per week
    number analyzed (Participants) | 31
    (all) | 15.4 (17.36)
Number of Participants According to Tobacco use [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set.
  Participants
    number analyzed (Participants) | 516
    Current Smoker | 38
    Previous Smoker | 88
    Never Smoked | 165
    Unknown | 225
Number of Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] — In this baseline characteristic number of cigarettes per day is reported in mean. Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Cigarettes per day
    For current smokers: number analyzed (Participants) | 32
    For current smokers | 20.4 (8.76)
    For previous smokers: number analyzed (Participants) | 58
    For previous smokers | 19.6 (13.27)
Number of Participants According to Source of Infection [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set.
  Participants
    number analyzed (Participants) | 516
    Hospital-acquired infections (HAI) | 354
    Healthcare-associated infections (HCAI) | 116
    Community-acquired infection (CAI) | 46
Number of Participants According to Other Indication for Ceftazidime-Avibactam [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Participants
    number analyzed (Participants) | 209
    Surgical site infection (SSI) | 15
    Central line associated blood stream infection (CLABSI) | 15
    Bloodstream infection (BSI)/ Sepsis | 97
    Meningitis | 0
    Endocarditis | 0
    Osteomyelitis | 7
    Febrile neutropenia | 24
    Other | 51
Number of Participants According to Initial Site of Infection [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Participants
    number analyzed (Participants) | 163
    Bladder | 2
    Kidney | 2
    Large Intestine | 5
    Lungs | 29
    Liver | 2
    Gall Bladder | 2
    Pancreas | 1
    Peritoneum | 4
    Small Intestine | 2
    Urethra | 11
    Other | 103
Number of Participants With Microbiological Cultures Performed for Current Infection Before Therapy [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the baseline characteristic.
  Participants
    number analyzed (Participants) | 239
    (all) | 239
Number of Pathogens Identified Before Ceftazidime-Avibactam Therapy [Number; unit: Pathogens] — Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Pathogens
    Gram-negative: Escherichia coli: number analyzed (Participants) | 239
    Gram-negative: Escherichia coli | 21
    Gram-negative: Klebsiella pneumoniae: number analyzed (Participants) | 239
    Gram-negative: Klebsiella pneumoniae | 140
    Gram-negative: Klebsiella species (spp): number analyzed (Participants) | 239
    Gram-negative: Klebsiella species (spp) | 25
    Gram-negative: Proteus mirabilis: number analyzed (Participants) | 239
    Gram-negative: Proteus mirabilis | 6
    Gram-negative: Proteus spp: number analyzed (Participants) | 239
    Gram-negative: Proteus spp | 1
    Gram-negative: Acinetobacter baumannii: number analyzed (Participants) | 239
    Gram-negative: Acinetobacter baumannii | 16
    Gram-negative: Acinetobacter spp: number analyzed (Participants) | 239
    Gram-negative: Acinetobacter spp | 1
    Gram-negative: Enterobacter cloacae: number analyzed (Participants) | 239
    Gram-negative: Enterobacter cloacae | 17
    Gram-negative: Enterobacter spp: number analyzed (Participants) | 239
    Gram-negative: Enterobacter spp | 5
    Gram-negative: Citrobacter spp: number analyzed (Participants) | 239
    Gram-negative: Citrobacter spp | 1
    Gram-negative: Serratia spp: number analyzed (Participants) | 239
    Gram-negative: Serratia spp | 3
    Gram-negative: Morganella morganii: number analyzed (Participants) | 239
    Gram-negative: Morganella morganii | 2
    Gram-negative: Pseudomonas aeruginosa: number analyzed (Participants) | 239
    Gram-negative: Pseudomonas aeruginosa | 30
    Gram-negative: Pseudomonas spp: number analyzed (Participants) | 239
    Gram-negative: Pseudomonas spp | 3
    Gram-negative: Haemophilus spp: number analyzed (Participants) | 239
    Gram-negative: Haemophilus spp | 1
    Gram-negative: Other: number analyzed (Participants) | 239
    Gram-negative: Other | 9
    Gram-positive: Staphylococcus aureus: number analyzed (Participants) | 239
    Gram-positive: Staphylococcus aureus | 7
    Gram-positive: Staphylococcus spp: number analyzed (Participants) | 239
    Gram-positive: Staphylococcus spp | 5
    Gram-positive: Enterococcus spp: number analyzed (Participants) | 239
    Gram-positive: Enterococcus spp | 23
    Gram-positive: Streptococcus spp: number analyzed (Participants) | 239
    Gram-positive: Streptococcus spp | 5
    Gram-positive: Other: number analyzed (Participants) | 239
    Gram-positive: Other | 10
    Anaerobes: Bacteroides spp: number analyzed (Participants) | 239
    Anaerobes: Bacteroides spp | 1
    Other Bacterial Agent: number analyzed (Participants) | 239
    Other Bacterial Agent | 3
Acute Physiology and Chronic Health Evaluation (APACHE) II Score [Mean (Standard Deviation); unit: Scores on a scale] — APACHE II assessed severity of illness in acutely ill participants. The point score was calculated from 12 admission physiologic variables comprising the Acute Physiology Score, the participants age, and chronic health status. The measurements computed for physiologic variables were transformed to integer APACHE II score ranging 0 (normal) to 71 (more severe). Higher scores indicate more severe disease and higher risk of death. Population: Data is presented for FAS72+ analysis set. Here, 'Number Analyzed' signifies number of participants evaluable for the baseline characteristic.
  Scores on a scale
    number analyzed (Participants) | 46
    (all) | 19.5 (7.93)
Number of Participants According to Indication for Ceftazidime-Avibactam [Count of Participants; unit: Participants] — Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Participants
    FAS72+: number analyzed (Participants) | 516
    FAS72+: Complicated Urinary Tract Infection (cUTI) | 103
    FAS72+: Complicated Intra-Abdominal Infection (cIAI) | 90
    FAS72+: Hospital-Acquired Pneumonia/Ventilator-Associated Pneumonia (HAP/VAP) | 114
    FAS72+: Other | 209
    FAS72-: number analyzed (Participants) | 53
    FAS72-: Complicated Urinary Tract Infection (cUTI) | 7
    FAS72-: Complicated Intra-Abdominal Infection (cIAI) | 12
    FAS72-: Hospital-Acquired Pneumonia/Ventilator-Associated Pneumonia (HAP/VAP) | 10
    FAS72-: Other | 24
Number of Participants With Comorbidities [Count of Participants; unit: Participants] — Population: Data is presented for FAS72+ analysis set.
  Participants
    number analyzed (Participants) | 516
    Any comorbidities | 479
    No comorbidities | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received at Least One Dose of Ceftazidime-Avibactam Classified According to Type of Usage as Monotherapy or Combination Therapy: FAS 72+ Population
Description: Number of participants who received at least one dose of ceftazidime-avibactam according to type of use as monotherapy or combination therapy was reported in this outcome measure. Index date was start date of ceftazidime-avibactam.
Time Frame: From start of index treatment to end of index treatment (maximum 179 days of treatment exposure) (from the data evaluated in approximately 40 months of the study)
Population: FAS72+ population included all participants with at least 72 hours of exposure to ceftazidime-avibactam.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants
  Monotherapy | 158
  Combination therapy | 358

2. Primary Outcome: Number of Participants Who Received at Least One Dose of Ceftazidime-Avibactam Classified According to Type of Usage as Monotherapy or Combination Therapy: FAS72- Population
Description: Number of participants who received at least one dose of ceftazidime-avibactam according to type of use as monotherapy or combination therapy was reported in this outcome measure.
Time Frame: From start of index treatment to end of index treatment (maximum 3 days of treatment exposure) (from the data evaluated in approximately 40 months of the study)
Population: FAS72- population included all participants with < 72 hours exposure to ceftazidime-avibactam. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 10
Participants
  Monotherapy | 3
  Combination therapy | 7

3. Primary Outcome: Total and Daily Dose of Ceftazidime-Avibactam: FAS72+ Population
Description: The total cumulative dose and daily dose of ceftazidime-avibactam was reported in this outcome measure. Total cumulative dose was defined as the sum of all doses received.
Time Frame: as for outcome 1
Population: FAS72+ population included all participants with at least 72 hours of exposure to ceftazidime-avibactam.
Measure: Mean (Standard Deviation); unit: Milligram (mg)
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Milligram (mg)
  Total dose | 62.2 (55.82)
  Daily dose | 5.2 (1.52)

4. Primary Outcome: Total and Daily Dose of Ceftazidime-Avibactam: FAS72- Population
Description: as for outcome 3
Time Frame: as for outcome 2
Population: FAS72- population included all participants with < 72 hours exposure to ceftazidime-avibactam.
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 53
Milligrams
  Total dose | 6.3 (3.65)
  Daily dose | 4.8 (1.96)

5. Primary Outcome: Number of Participants Classified According to Frequency of Dosing: FAS72+ Population
Description: Number of participants classified according to frequency of dose (once daily [OD], every other day [QOD], post-dialysis, each 48 hours [h], three times daily [TID], twice daily [BD], four times daily [QID], once loading dose [an initial higher dose of a drug that may be given at the beginning of a course of treatment before dropping down to a lower maintenance dose], every three days, once, etc.,) for ceftazidime-avibactam were reported in this outcome measure.
Time Frame: as for outcome 1
Population: FAS72+ population included all participants with at least 72 hours of exposure to ceftazidime-avibactam.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants
  0.75 grams (g)*OD | 4
  0.75 g*QOD | 4
  0.75 g*Other: Post dialysis | 1
  0.75 g*Other: each 48 h | 1
  0.75 g*TID | 1
  0.75 g*BD | 13
  0.80 g*BD | 2
  0.94 g*BD | 1
  1.00 g*OD | 6
  1.00 g*QOD | 2
  1.00 g*QID | 2
  1.00 g*Other: Post dialysis | 1
  1.00 g*TID | 51
  1.00 g*BD | 19
  1.20 g*TID | 1
  1.25 g*TID | 1
  1.50 g*OD | 1
  2.00 g*OD | 7
  2.00 g*QOD | 2
  2.00 g*QID | 5
  2.00 g*Other: Once, loading dose | 2
  2.00 g*Other: every 3 days | 1
  2.00 g*Other: once | 1
  2.00 g*TID | 400
  2.00 g*BD | 29
  2.50 g*OD | 1

6. Primary Outcome: Number of Participants Classified According to Frequency of Dosing: FAS72- Population
Description: Number of participants classified according to frequency of dose (once daily [OD], every other day [QOD], each 48 hours [h], continuous infusion per 48 hours [c/48 h], three times daily [TID], twice daily [BD], four times daily [QID], one dose, loading dose [an initial higher dose of a drug that may be given at the beginning of a course of treatment before dropping down to a lower maintenance dose] etc.,) for ceftazidime-avibactam were reported in this outcome measure.
Time Frame: as for outcome 2
Population: FAS72- population included all participants with < 72 hours exposure to ceftazidime-avibactam.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 53
Participants
  0.75 g*Other: 48 h | 1
  0.94 g*QOD | 1
  1.00 g*OD | 2
  1.00 g*QOD | 1
  1.00 g*Other: 48 h | 1
  1.00 g*Other: c/48h | 1
  1.00 g*TID | 3
  1.87 g*BD | 1
  2.00 g*OD | 3
  2.00 g*QID | 1
  2.00 g*Other: Loading dose | 1
  2.00 g*Other: one dose | 1
  2.00 g*TID | 34
  2.00 g*BD | 4
  3.00 g*BD | 1

7. Primary Outcome: Total Duration of Administration of Ceftazidime-Avibactam: FAS72+ Population
Description: Total duration of administration was calculated as stop date of administration of ceftazidime-avibactam minus start date of ceftazidime-avibactam administration plus 1.
Time Frame: as for outcome 1
Population: FAS72+ population included all participants with at least 72 hours of exposure to ceftazidime-avibactam.
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Days | 9.0 [2 to 179]

8. Primary Outcome: Total Duration of Administration of Ceftazidime-Avibactam: FAS72- Population
Description: as for outcome 7
Time Frame: as for outcome 2
Population: FAS72- population included all participants with < 72 hours exposure to ceftazidime-avibactam.
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 53
Days | 1.0 [1 to 3]

9. Primary Outcome: Number of Participants Classified According to Reason for Discontinuation of Ceftazidime-Avibactam: FAS72+ Population
Description: Number of participants according to the reasons for discontinuation of ceftazidime-avibactam were reported in this outcome measure.
Time Frame: as for outcome 1
Population: FAS72+ population included all participants with at least 72 hours of exposure to ceftazidime-avibactam. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 506
Participants
  Adverse events (AEs) | 3
  Perceived clinical failure/disease progression | 10
  Isolation of a resistant pathogen | 9
  Preference for empiric coverage | 2
  Secondary infection requiring regimen change | 11
  Switch to oral therapy | 5
  De-escalation | 59
  Cure | 329
  Death | 50
  Other | 28

10. Primary Outcome: Number of Participants Classified According to Reason for Discontinuation of Ceftazidime-Avibactam: FAS72- Population
Description: as for outcome 9
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 52
Participants
  Adverse events (AEs) | 0
  Perceived clinical failure/disease progression | 1
  Isolation of a resistant pathogen | 6
  Preference for empiric coverage | 1
  Secondary infection requiring regimen change | 2
  Switch to oral therapy | 0
  De-escalation | 23
  Cure | 1
  Death | 14
  Other | 4

11. Primary Outcome: Number of Participants Classified According to Antibiotics Used Concurrently: FAS 72+ Population
Description: The number of participants classified according to antibiotics used concurrently with ceftazidime-avibactam were reported in this outcome measure. Participants could have received more than 1 antibiotic.
Time Frame: as for outcome 1
Population: FAS72+ population included all participants with at least 72 hours of exposure to Ceftazidime-avibactam.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants
  Aminoglycoside: Amikacin | 58
  Aminoglycoside: Gentamicin | 19
  Aminoglycoside: Tobramycin | 6
  Amphenicol: Chloramphenicol | 1
  Carbapenems: Doripenem | 1
  Carbapenems: Ertapenem | 1
  Carbapenems: Imipenem | 1
  Carbapenems: Meropenem | 28
  Cephalosporins: Ceftazidime | 4
  Glycopeptides: Teicoplanin | 18
  Glycopeptides: Telavancin | 1
  Glycopeptides: Vancomycin | 65
  Glycylcycline: Tigecycline | 49
  Lipopeptides: Daptomycin | 21
  Macrolides: Azithromycin | 4
  Macrolides: Clarithromycin | 2
  Macrolides: Clindamycin | 1
  Macrolides: Erythromycin | 6
  Macrolides: Fidaxomicin | 1
  Monobactam: Aztreonam | 104
  Nitroimidazole: Metronidazole | 60
  Oxazolidinones: Linezolid | 37
  Oxazolidinones: Tedizolid | 4
  Penicillins: Amoxicillin | 1
  Penicillins: Ampicillin | 8
  Penicillins: Benzylpenicillin | 1
  Penicillins: Flucloxacillin | 1
  Penicillins: Ticarcillin | 1
  Penicillins and beta-lactamase inhibitors: Amoxicillin-clavulanate | 1
  Penicillins and beta-lactamase inhibitors: Ampicillin-sulbactam | 1
  Penicillins and beta-lactamase inhibitors: Piperacillin-tazobactam | 5
  Fluoroquinolones: Ciprofloxacin | 15
  Fluoroquinolones: Levofloxacin | 5
  Fluoroquinolones: Moxifloxacin | 3
  Fluoroquinolones: Ofloxacin ear drops | 1
  Tetracycline: Doxycycline | 1
  Other agents | 123
  Polymyxins: Colistin | 60
  Polymyxins: Polymyxin B | 15
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole | 21
  Other antibiotics: Clofazimine | 1
  Other antibiotics: Ethambutol | 1
  Other antibiotics: Fosfomycin | 12
  Other antibiotics: Isoniazid | 2
  Other antibiotics: Rifampicin | 1
  Other antibiotics: Rifaximin | 1

12. Primary Outcome: Number of Participants Classified According to Reason for Initiating Antibiotics: FAS 72+ Population
Description: The number of participants classified according to reason for initiating specific antibiotics combined with ceftazidime-avibactam were reported in this outcome measure. One participant could have received more than 1 antibiotics and there could be more than 1 reason for initiating antibiotics.
Time Frame: as for outcome 1
Population: FAS72+ population included all participants with at least 72 hours of exposure to ceftazidime-avibactam. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants
  Amikacin: Empiric treatment: number analyzed (Participants) | 58
  Amikacin: Empiric treatment | 7
  Amikacin: Failure of antimicrobial treatment: number analyzed (Participants) | 58
  Amikacin: Failure of antimicrobial treatment | 2
  Amikacin: Infection: number analyzed (Participants) | 58
  Amikacin: Infection | 30
  Amikacin: Microbiology: number analyzed (Participants) | 58
  Amikacin: Microbiology | 18
  Amikacin: Prophylaxis: number analyzed (Participants) | 58
  Amikacin: Prophylaxis | 1
  Amikacin: Other: number analyzed (Participants) | 58
  Amikacin: Other | 1
  Amoxicillin: Microbiology: number analyzed (Participants) | 1
  Amoxicillin: Microbiology | 1
  Amoxicillin-clavulanate: Microbiology: number analyzed (Participants) | 1
  Amoxicillin-clavulanate: Microbiology | 1
  Ampicillin: Infection: number analyzed (Participants) | 8
  Ampicillin: Infection | 3
  Ampicillin: Microbiology: number analyzed (Participants) | 8
  Ampicillin: Microbiology | 4
  Ampicillin: Other: number analyzed (Participants) | 8
  Ampicillin: Other | 1
  Ampicillin-sulbactam: Infection: number analyzed (Participants) | 1
  Ampicillin-sulbactam: Infection | 1
  Aztreonam: Disease progression: number analyzed (Participants) | 102
  Aztreonam: Disease progression | 1
  Aztreonam: Empiric treatment: number analyzed (Participants) | 102
  Aztreonam: Empiric treatment | 1
  Aztreonam: Failure of antimicrobial treatment: number analyzed (Participants) | 102
  Aztreonam: Failure of antimicrobial treatment | 4
  Aztreonam: Infection: number analyzed (Participants) | 102
  Aztreonam: Infection | 23
  Aztreonam: Microbiology: number analyzed (Participants) | 102
  Aztreonam: Microbiology | 73
  Aztreonam: Other: number analyzed (Participants) | 102
  Aztreonam: Other | 1
  Ceftazidime: Infection: number analyzed (Participants) | 4
  Ceftazidime: Infection | 2
  Ceftazidime: Microbiology: number analyzed (Participants) | 4
  Ceftazidime: Microbiology | 2
  Chloramphenicol: Infection: number analyzed (Participants) | 1
  Chloramphenicol: Infection | 1
  Ciprofloxacin: Infection: number analyzed (Participants) | 15
  Ciprofloxacin: Infection | 8
  Ciprofloxacin: Microbiology: number analyzed (Participants) | 15
  Ciprofloxacin: Microbiology | 6
  Ciprofloxacin: Prophylaxis: number analyzed (Participants) | 15
  Ciprofloxacin: Prophylaxis | 1
  Doripenem: Infection: number analyzed (Participants) | 1
  Doripenem: Infection | 1
  Ertapenem: Microbiology: number analyzed (Participants) | 1
  Ertapenem: Microbiology | 1
  Gentamicin: Empiric treatment: number analyzed (Participants) | 19
  Gentamicin: Empiric treatment | 2
  Gentamicin: Infection: number analyzed (Participants) | 19
  Gentamicin: Infection | 5
  Gentamicin: Microbiology: number analyzed (Participants) | 19
  Gentamicin: Microbiology | 13
  Imipenem: Empiric treatment: number analyzed (Participants) | 1
  Imipenem: Empiric treatment | 1
  Levofloxacin: Infection: number analyzed (Participants) | 5
  Levofloxacin: Infection | 3
  Levofloxacin: Microbiology: number analyzed (Participants) | 5
  Levofloxacin: Microbiology | 2
  Meropenem: Empiric treatment: number analyzed (Participants) | 28
  Meropenem: Empiric treatment | 3
  Meropenem: Infection: number analyzed (Participants) | 28
  Meropenem: Infection | 14
  Meropenem: Microbiology: number analyzed (Participants) | 28
  Meropenem: Microbiology | 9
  Meropenem: Prophylaxis: number analyzed (Participants) | 28
  Meropenem: Prophylaxis | 1
  Meropenem: Other: number analyzed (Participants) | 28
  Meropenem: Other | 2
  Moxifloxacin: Infection: number analyzed (Participants) | 3
  Moxifloxacin: Infection | 2
  Moxifloxacin: Microbiology: number analyzed (Participants) | 3
  Moxifloxacin: Microbiology | 1
  Piperacillin-tazobactam: Empiric treatment: number analyzed (Participants) | 4
  Piperacillin-tazobactam: Empiric treatment | 1
  Piperacillin-tazobactam: Infection: number analyzed (Participants) | 4
  Piperacillin-tazobactam: Infection | 1
  Piperacillin-tazobactam: Microbiology: number analyzed (Participants) | 4
  Piperacillin-tazobactam: Microbiology | 2
  Ticarcillin: Infection: number analyzed (Participants) | 1
  Ticarcillin: Infection | 1
  Tigecycline: Disease progression: number analyzed (Participants) | 48
  Tigecycline: Disease progression | 1
  Tigecycline: Empiric treatment: number analyzed (Participants) | 48
  Tigecycline: Empiric treatment | 1
  Tigecycline: Failure of antimicrobial treatment: number analyzed (Participants) | 48
  Tigecycline: Failure of antimicrobial treatment | 2
  Tigecycline: Infection: number analyzed (Participants) | 48
  Tigecycline: Infection | 21
  Tigecycline: Microbiology: number analyzed (Participants) | 48
  Tigecycline: Microbiology | 20
  Tigecycline: Other: number analyzed (Participants) | 48
  Tigecycline: Other | 3
  Tobramycin: Infection: number analyzed (Participants) | 6
  Tobramycin: Infection | 5
  Tobramycin: Other: number analyzed (Participants) | 6
  Tobramycin: Other | 1
  Polymyxins: Colistin: Disease progression: number analyzed (Participants) | 59
  Polymyxins: Colistin: Disease progression | 1
  Polymyxins: Colistin: Empiric treatment: number analyzed (Participants) | 59
  Polymyxins: Colistin: Empiric treatment | 1
  Polymyxins: Colistin: Infection: number analyzed (Participants) | 59
  Polymyxins: Colistin: Infection | 30
  Polymyxins: Colistin: Microbiology: number analyzed (Participants) | 59
  Polymyxins: Colistin: Microbiology | 27
  Polymyxins: Colistin: Other: number analyzed (Participants) | 59
  Polymyxins: Colistin: Other | 2
  Polymyxins: Polymyxin B: Infection: number analyzed (Participants) | 15
  Polymyxins: Polymyxin B: Infection | 6
  Polymyxins: Polymyxin B: Microbiology: number analyzed (Participants) | 15
  Polymyxins: Polymyxin B: Microbiology | 9
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Disease progression: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Disease progression | 1
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Empiric treatment: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Empiric treatment | 1
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Failure of antimicrobial treatment: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Failure of antimicrobial treatment | 1
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Infection: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Infection | 5
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Microbiology: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Microbiology | 8
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Prophylaxis: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Prophylaxis | 5
  Other antibiotics: Fosfomycin: Disease progression: number analyzed (Participants) | 11
  Other antibiotics: Fosfomycin: Disease progression | 1
  Other antibiotics: Fosfomycin: Infection: number analyzed (Participants) | 11
  Other antibiotics: Fosfomycin: Infection | 1
  Other antibiotics: Fosfomycin: Microbiology: number analyzed (Participants) | 11
  Other antibiotics: Fosfomycin: Microbiology | 8
  Other antibiotics: Fosfomycin: Other: number analyzed (Participants) | 11
  Other antibiotics: Fosfomycin: Other | 1
  Other antibiotics: Rifampicin: Microbiology: number analyzed (Participants) | 1
  Other antibiotics: Rifampicin: Microbiology | 1
  Azithromycin: Infection: number analyzed (Participants) | 4
  Azithromycin: Infection | 2
  Azithromycin: Microbiology: number analyzed (Participants) | 4
  Azithromycin: Microbiology | 1
  Azithromycin: Other: number analyzed (Participants) | 4
  Azithromycin: Other | 1
  Benzylpenicillin: Microbiology: number analyzed (Participants) | 1
  Benzylpenicillin: Microbiology | 1
  Clarithromycin: Microbiology: number analyzed (Participants) | 2
  Clarithromycin: Microbiology | 2
  Clindamycin: Empiric treatment: number analyzed (Participants) | 1
  Clindamycin: Empiric treatment | 1
  Daptomycin: Empiric treatment: number analyzed (Participants) | 21
  Daptomycin: Empiric treatment | 1
  Daptomycin: Infection: number analyzed (Participants) | 21
  Daptomycin: Infection | 16
  Daptomycin: Microbiology: number analyzed (Participants) | 21
  Daptomycin: Microbiology | 2
  Daptomycin: Other: number analyzed (Participants) | 21
  Daptomycin: Other | 2
  Doxycycline: Infection: number analyzed (Participants) | 1
  Doxycycline: Infection | 1
  Erythromycin: Infection: number analyzed (Participants) | 6
  Erythromycin: Infection | 2
  Erythromycin: Other: number analyzed (Participants) | 6
  Erythromycin: Other | 4
  Fidaxomicin: Clostridium difficile: number analyzed (Participants) | 1
  Fidaxomicin: Clostridium difficile | 1
  Flucloxacillin: Infection: number analyzed (Participants) | 1
  Flucloxacillin: Infection | 1
  Linezolid: Disease progression: number analyzed (Participants) | 37
  Linezolid: Disease progression | 1
  Linezolid: Empiric treatment: number analyzed (Participants) | 37
  Linezolid: Empiric treatment | 6
  Linezolid: Failure of antimicrobial treatment: number analyzed (Participants) | 37
  Linezolid: Failure of antimicrobial treatment | 2
  Linezolid: Infection: number analyzed (Participants) | 37
  Linezolid: Infection | 15
  Linezolid: Microbiology: number analyzed (Participants) | 37
  Linezolid: Microbiology | 13
  Tedizolid: Infection: number analyzed (Participants) | 4
  Tedizolid: Infection | 2
  Tedizolid: Microbiology: number analyzed (Participants) | 4
  Tedizolid: Microbiology | 2
  Teicoplanin: Clostridium difficile: number analyzed (Participants) | 17
  Teicoplanin: Clostridium difficile | 1
  Teicoplanin: Disease progression: number analyzed (Participants) | 17
  Teicoplanin: Disease progression | 1
  Teicoplanin: Empiric treatment: number analyzed (Participants) | 17
  Teicoplanin: Empiric treatment | 2
  Teicoplanin: Infection: number analyzed (Participants) | 17
  Teicoplanin: Infection | 4
  Teicoplanin: Microbiology: number analyzed (Participants) | 17
  Teicoplanin: Microbiology | 7
  Teicoplanin: Prophylaxis: number analyzed (Participants) | 17
  Teicoplanin: Prophylaxis | 2
  Telavancin: Disease progression: number analyzed (Participants) | 1
  Telavancin: Disease progression | 1
  Vancomycin: Clostridium difficile: number analyzed (Participants) | 65
  Vancomycin: Clostridium difficile | 6
  Vancomycin: Empiric treatment: number analyzed (Participants) | 65
  Vancomycin: Empiric treatment | 2
  Vancomycin: Infection: number analyzed (Participants) | 65
  Vancomycin: Infection | 40
  Vancomycin: Microbiology: number analyzed (Participants) | 65
  Vancomycin: Microbiology | 14
  Vancomycin: Prophylaxis: number analyzed (Participants) | 65
  Vancomycin: Prophylaxis | 3
  Vancomycin: Other: number analyzed (Participants) | 65
  Vancomycin: Other | 2
  Other antibiotics: Rifaximin: Infection: number analyzed (Participants) | 1
  Other antibiotics: Rifaximin: Infection | 1
  Metronidazole: Clostridium difficile: number analyzed (Participants) | 59
  Metronidazole: Clostridium difficile | 9
  Metronidazole: Empiric treatment: number analyzed (Participants) | 59
  Metronidazole: Empiric treatment | 2
  Metronidazole: Failure of antimicrobial treatment: number analyzed (Participants) | 59
  Metronidazole: Failure of antimicrobial treatment | 2
  Metronidazole: Infection: number analyzed (Participants) | 59
  Metronidazole: Infection | 28
  Metronidazole: Microbiology: number analyzed (Participants) | 59
  Metronidazole: Microbiology | 18
  Metronidazole: Prophylaxis: number analyzed (Participants) | 59
  Metronidazole: Prophylaxis | 1
  Metronidazole: Other: number analyzed (Participants) | 59
  Metronidazole: Other | 3
  Ofloxacin ear drops: Infection: number analyzed (Participants) | 1
  Ofloxacin ear drops: Infection | 1
  Other antibiotics: Clofazimine: Infection: number analyzed (Participants) | 1
  Other antibiotics: Clofazimine: Infection | 1
  Ethambutol: Microbiology: number analyzed (Participants) | 1
  Ethambutol: Microbiology | 1
  Isoniazid: Microbiology: number analyzed (Participants) | 2
  Isoniazid: Microbiology | 1
  Isoniazid: Prophylaxis: number analyzed (Participants) | 2
  Isoniazid: Prophylaxis | 1

13. Primary Outcome: Number of Participants Classified According to Reason for Discontinuing Antibiotics: FAS 72+ Population
Description: The number of participants classified according to reason for discontinuing specific antibiotics combined with ceftazidime-avibactam were reported in this outcome measure. One participant could have received more than 1 antibiotics and there could be more than 1 reason for discontinuing antibiotics.
Time Frame: as for outcome 1
Population: FAS72+ population included all participants with at least 72 hours of exposure to Ceftazidime-avibactam. Here, "Number Analyzed" signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants
  Amikacin: Perceived clinical failure/disease progression: number analyzed (Participants) | 58
  Amikacin: Perceived clinical failure/disease progression | 4
  Amikacin: Isolation of a resistant pathogen: number analyzed (Participants) | 58
  Amikacin: Isolation of a resistant pathogen | 5
  Amikacin: Preference for empiric coverage: number analyzed (Participants) | 58
  Amikacin: Preference for empiric coverage | 6
  Amikacin: Secondary infection requiring regimen change: number analyzed (Participants) | 58
  Amikacin: Secondary infection requiring regimen change | 1
  Amikacin: De-escalation: number analyzed (Participants) | 58
  Amikacin: De-escalation | 13
  Amikacin: Cure: number analyzed (Participants) | 58
  Amikacin: Cure | 15
  Amikacin: Death: number analyzed (Participants) | 58
  Amikacin: Death | 1
  Amikacin: Other: number analyzed (Participants) | 58
  Amikacin: Other | 15
  Amoxicillin: Cure: number analyzed (Participants) | 1
  Amoxicillin: Cure | 1
  Amoxicillin-clavulanate: Cure: number analyzed (Participants) | 1
  Amoxicillin-clavulanate: Cure | 1
  Ampicillin: Switch to oral therapy: number analyzed (Participants) | 7
  Ampicillin: Switch to oral therapy | 1
  Ampicillin: Cure: number analyzed (Participants) | 7
  Ampicillin: Cure | 6
  Ampicillin: Other: number analyzed (Participants) | 7
  Ampicillin: Other | 1
  Ampicillin-sulbactam: De-escalation: number analyzed (Participants) | 1
  Ampicillin-sulbactam: De-escalation | 1
  Aztreonam: Perceived clinical failure/disease progression: number analyzed (Participants) | 98
  Aztreonam: Perceived clinical failure/disease progression | 3
  Aztreonam: Isolation of a resistant pathogen: number analyzed (Participants) | 98
  Aztreonam: Isolation of a resistant pathogen | 3
  Aztreonam: Preference for empiric coverage: number analyzed (Participants) | 98
  Aztreonam: Preference for empiric coverage | 2
  Aztreonam: Secondary infection requiring regimen change: number analyzed (Participants) | 98
  Aztreonam: Secondary infection requiring regimen change | 1
  Aztreonam: Switch to oral therapy: number analyzed (Participants) | 98
  Aztreonam: Switch to oral therapy | 2
  Aztreonam: De-escalation: number analyzed (Participants) | 98
  Aztreonam: De-escalation | 11
  Aztreonam: Cure: number analyzed (Participants) | 98
  Aztreonam: Cure | 66
  Aztreonam: Death: number analyzed (Participants) | 98
  Aztreonam: Death | 11
  Aztreonam: Other: number analyzed (Participants) | 98
  Aztreonam: Other | 2
  Ceftazidime: De-escalation: number analyzed (Participants) | 4
  Ceftazidime: De-escalation | 1
  Ceftazidime: Cure: number analyzed (Participants) | 4
  Ceftazidime: Cure | 1
  Ceftazidime: Death: number analyzed (Participants) | 4
  Ceftazidime: Death | 1
  Ceftazidime: Other: number analyzed (Participants) | 4
  Ceftazidime: Other | 1
  Chloramphenicol: Cure: number analyzed (Participants) | 1
  Chloramphenicol: Cure | 1
  Ciprofloxacin: Perceived clinical failure/disease progression: number analyzed (Participants) | 15
  Ciprofloxacin: Perceived clinical failure/disease progression | 1
  Ciprofloxacin: Isolation of a resistant pathogen: number analyzed (Participants) | 15
  Ciprofloxacin: Isolation of a resistant pathogen | 1
  Ciprofloxacin: Preference for empiric coverage: number analyzed (Participants) | 15
  Ciprofloxacin: Preference for empiric coverage | 1
  Ciprofloxacin: Switch to oral therapy: number analyzed (Participants) | 15
  Ciprofloxacin: Switch to oral therapy | 1
  Ciprofloxacin: De-escalation: number analyzed (Participants) | 15
  Ciprofloxacin: De-escalation | 3
  Ciprofloxacin: Cure: number analyzed (Participants) | 15
  Ciprofloxacin: Cure | 4
  Ciprofloxacin: Death: number analyzed (Participants) | 15
  Ciprofloxacin: Death | 2
  Ciprofloxacin: Other: number analyzed (Participants) | 15
  Ciprofloxacin: Other | 3
  Doripenem: Cure: number analyzed (Participants) | 1
  Doripenem: Cure | 1
  Ertapenem: Cure: number analyzed (Participants) | 1
  Ertapenem: Cure | 1
  Gentamicin: Isolation of a resistant pathogen: number analyzed (Participants) | 19
  Gentamicin: Isolation of a resistant pathogen | 4
  Gentamicin: Preference for empiric coverage: number analyzed (Participants) | 19
  Gentamicin: Preference for empiric coverage | 3
  Gentamicin: De-escalation: number analyzed (Participants) | 19
  Gentamicin: De-escalation | 4
  Gentamicin: Cure: number analyzed (Participants) | 19
  Gentamicin: Cure | 5
  Gentamicin: Other: number analyzed (Participants) | 19
  Gentamicin: Other | 4
  Imipenem: Secondary infection requiring regimen change: number analyzed (Participants) | 1
  Imipenem: Secondary infection requiring regimen change | 1
  Levofloxacin: Perceived clinical failure/disease progression: number analyzed (Participants) | 5
  Levofloxacin: Perceived clinical failure/disease progression | 1
  Levofloxacin: Secondary infection requiring regimen change: number analyzed (Participants) | 5
  Levofloxacin: Secondary infection requiring regimen change | 1
  Levofloxacin: De-escalation: number analyzed (Participants) | 5
  Levofloxacin: De-escalation | 1
  Levofloxacin: Death: number analyzed (Participants) | 5
  Levofloxacin: Death | 1
  Levofloxacin: Other: number analyzed (Participants) | 5
  Levofloxacin: Other | 1
  Meropenem: AE: number analyzed (Participants) | 28
  Meropenem: AE | 1
  Meropenem: Perceived clinical failure/disease progression: number analyzed (Participants) | 28
  Meropenem: Perceived clinical failure/disease progression | 3
  Meropenem: Isolation of a resistant pathogen: number analyzed (Participants) | 28
  Meropenem: Isolation of a resistant pathogen | 5
  Meropenem: Preference for empiric coverage: number analyzed (Participants) | 28
  Meropenem: Preference for empiric coverage | 3
  Meropenem: Secondary infection requiring regimen change: number analyzed (Participants) | 28
  Meropenem: Secondary infection requiring regimen change | 1
  Meropenem: Switch to oral therapy: number analyzed (Participants) | 28
  Meropenem: Switch to oral therapy | 1
  Meropenem: De-escalation: number analyzed (Participants) | 28
  Meropenem: De-escalation | 6
  Meropenem: Cure: number analyzed (Participants) | 28
  Meropenem: Cure | 5
  Meropenem: Death: number analyzed (Participants) | 28
  Meropenem: Death | 2
  Meropenem: Other: number analyzed (Participants) | 28
  Meropenem: Other | 3
  Moxifloxacin: Switch to oral therapy: number analyzed (Participants) | 3
  Moxifloxacin: Switch to oral therapy | 1
  Moxifloxacin: Cure: number analyzed (Participants) | 3
  Moxifloxacin: Cure | 1
  Moxifloxacin: Other: number analyzed (Participants) | 3
  Moxifloxacin: Other | 1
  Piperacillin-tazobactam: Preference for empiric coverage: number analyzed (Participants) | 4
  Piperacillin-tazobactam: Preference for empiric coverage | 1
  Piperacillin-tazobactam: Secondary infection requiring regimen change: number analyzed (Participants) | 4
  Piperacillin-tazobactam: Secondary infection requiring regimen change | 1
  Piperacillin-tazobactam: De-escalation: number analyzed (Participants) | 4
  Piperacillin-tazobactam: De-escalation | 1
  Piperacillin-tazobactam: Cure: number analyzed (Participants) | 4
  Piperacillin-tazobactam: Cure | 1
  Ticarcillin: Cure: number analyzed (Participants) | 1
  Ticarcillin: Cure | 1
  Tigecycline: AE: number analyzed (Participants) | 48
  Tigecycline: AE | 1
  Tigecycline: Perceived clinical failure/disease progression: number analyzed (Participants) | 48
  Tigecycline: Perceived clinical failure/disease progression | 4
  Tigecycline: Isolation of a resistant pathogen: number analyzed (Participants) | 48
  Tigecycline: Isolation of a resistant pathogen | 3
  Tigecycline: De-escalation: number analyzed (Participants) | 48
  Tigecycline: De-escalation | 8
  Tigecycline: Cure: number analyzed (Participants) | 48
  Tigecycline: Cure | 23
  Tigecycline: Death: number analyzed (Participants) | 48
  Tigecycline: Death | 9
  Tigecycline: Other: number analyzed (Participants) | 48
  Tigecycline: Other | 5
  Tobramycin: Preference for empiric coverage: number analyzed (Participants) | 6
  Tobramycin: Preference for empiric coverage | 1
  Tobramycin: Secondary infection requiring regimen change: number analyzed (Participants) | 6
  Tobramycin: Secondary infection requiring regimen change | 1
  Tobramycin: Cure: number analyzed (Participants) | 6
  Tobramycin: Cure | 3
  Tobramycin: Other: number analyzed (Participants) | 6
  Tobramycin: Other | 1
  Polymyxins: Colistin: AE: number analyzed (Participants) | 58
  Polymyxins: Colistin: AE | 3
  Polymyxins: Colistin: Perceived clinical failure/disease progression: number analyzed (Participants) | 58
  Polymyxins: Colistin: Perceived clinical failure/disease progression | 2
  Polymyxins: Colistin: Isolation of a resistant pathogen: number analyzed (Participants) | 58
  Polymyxins: Colistin: Isolation of a resistant pathogen | 6
  Polymyxins: Colistin: Preference for empiric coverage: number analyzed (Participants) | 58
  Polymyxins: Colistin: Preference for empiric coverage | 2
  Polymyxins: Colistin: De-escalation: number analyzed (Participants) | 58
  Polymyxins: Colistin: De-escalation | 15
  Polymyxins: Colistin: Cure: number analyzed (Participants) | 58
  Polymyxins: Colistin: Cure | 19
  Polymyxins: Colistin: Death: number analyzed (Participants) | 58
  Polymyxins: Colistin: Death | 11
  Polymyxins: Colistin: Other: number analyzed (Participants) | 58
  Polymyxins: Colistin: Other | 5
  Polymyxins: Polymyxin B: Perceived clinical failure/disease progression: number analyzed (Participants) | 15
  Polymyxins: Polymyxin B: Perceived clinical failure/disease progression | 1
  Polymyxins: Polymyxin B: Isolation of a resistant pathogen: number analyzed (Participants) | 15
  Polymyxins: Polymyxin B: Isolation of a resistant pathogen | 1
  Polymyxins: Polymyxin B: De-escalation: number analyzed (Participants) | 15
  Polymyxins: Polymyxin B: De-escalation | 6
  Polymyxins: Polymyxin B: Cure: number analyzed (Participants) | 15
  Polymyxins: Polymyxin B: Cure | 4
  Polymyxins: Polymyxin B: Death: number analyzed (Participants) | 15
  Polymyxins: Polymyxin B: Death | 2
  Polymyxins: Polymyxin B: Other: number analyzed (Participants) | 15
  Polymyxins: Polymyxin B: Other | 1
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole (sulfa) : AE: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole (sulfa) : AE | 3
  Sulfonamides and Trimethoprim: Trimethoprim-sulfa: Perceived clinical failure/disease progression: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfa: Perceived clinical failure/disease progression | 1
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Preference for empiric coverage: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Preference for empiric coverage | 2
  Sulfonamides and Trimethoprim: Trimethoprim-sulfa: Secondary infection requiring regimen change: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfa: Secondary infection requiring regimen change | 1
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: De-escalation: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: De-escalation | 2
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Cure: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Cure | 7
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Death: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Death | 2
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Other: number analyzed (Participants) | 20
  Sulfonamides and Trimethoprim: Trimethoprim-sulfamethoxazole: Other | 3
  Fosfomycin: Perceived clinical failure/disease progression: number analyzed (Participants) | 10
  Fosfomycin: Perceived clinical failure/disease progression | 1
  Fosfomycin: Isolation of a resistant pathogen: number analyzed (Participants) | 10
  Fosfomycin: Isolation of a resistant pathogen | 1
  Fosfomycin: De-escalation: number analyzed (Participants) | 10
  Fosfomycin: De-escalation | 1
  Fosfomycin: Cure: number analyzed (Participants) | 10
  Fosfomycin: Cure | 5
  Fosfomycin: Death: number analyzed (Participants) | 10
  Fosfomycin: Death | 2
  Rifampicin: Other: number analyzed (Participants) | 1
  Rifampicin: Other | 1
  Azithromycin: Perceived clinical failure/disease progression: number analyzed (Participants) | 4
  Azithromycin: Perceived clinical failure/disease progression | 1
  Azithromycin: Preference for empiric coverage: number analyzed (Participants) | 4
  Azithromycin: Preference for empiric coverage | 1
  Azithromycin: Other: number analyzed (Participants) | 4
  Azithromycin: Other | 2
  Benzylpenicillin: Cure: number analyzed (Participants) | 1
  Benzylpenicillin: Cure | 1
  Clarithromycin: De-escalation: number analyzed (Participants) | 2
  Clarithromycin: De-escalation | 1
  Clarithromycin: Cure: number analyzed (Participants) | 2
  Clarithromycin: Cure | 1
  Clindamycin: Preference for empiric coverage: number analyzed (Participants) | 1
  Clindamycin: Preference for empiric coverage | 1
  Daptomycin: AE: number analyzed (Participants) | 21
  Daptomycin: AE | 1
  Daptomycin: Perceived clinical failure/disease progression: number analyzed (Participants) | 21
  Daptomycin: Perceived clinical failure/disease progression | 1
  Daptomycin: Isolation of a resistant pathogen: number analyzed (Participants) | 21
  Daptomycin: Isolation of a resistant pathogen | 4
  Daptomycin: Switch to oral therapy: number analyzed (Participants) | 21
  Daptomycin: Switch to oral therapy | 1
  Daptomycin: De-escalation: number analyzed (Participants) | 21
  Daptomycin: De-escalation | 5
  Daptomycin: Cure: number analyzed (Participants) | 21
  Daptomycin: Cure | 5
  Daptomycin: Death: number analyzed (Participants) | 21
  Daptomycin: Death | 2
  Daptomycin: Other: number analyzed (Participants) | 21
  Daptomycin: Other | 3
  Doxycycline: Other: number analyzed (Participants) | 1
  Doxycycline: Other | 1
  Erythromycin: De-escalation: number analyzed (Participants) | 6
  Erythromycin: De-escalation | 1
  Erythromycin: Cure: number analyzed (Participants) | 6
  Erythromycin: Cure | 2
  Erythromycin: Death: number analyzed (Participants) | 6
  Erythromycin: Death | 1
  Erythromycin: Other: number analyzed (Participants) | 6
  Erythromycin: Other | 2
  Fidaxomicin: Cure: number analyzed (Participants) | 1
  Fidaxomicin: Cure | 1
  Flucloxacillin: Preference for empiric coverage: number analyzed (Participants) | 1
  Flucloxacillin: Preference for empiric coverage | 1
  Linezolid: AE: number analyzed (Participants) | 36
  Linezolid: AE | 1
  Linezolid: Perceived clinical failure/disease progression: number analyzed (Participants) | 36
  Linezolid: Perceived clinical failure/disease progression | 1
  Linezolid: Isolation of a resistant pathogen: number analyzed (Participants) | 36
  Linezolid: Isolation of a resistant pathogen | 1
  Linezolid: Preference for empiric coverage: number analyzed (Participants) | 36
  Linezolid: Preference for empiric coverage | 1
  Linezolid: Secondary infection requiring regimen change: number analyzed (Participants) | 36
  Linezolid: Secondary infection requiring regimen change | 2
  Linezolid: Switch to oral therapy: number analyzed (Participants) | 36
  Linezolid: Switch to oral therapy | 2
  Linezolid: De-escalation: number analyzed (Participants) | 36
  Linezolid: De-escalation | 4
  Linezolid: Cure: number analyzed (Participants) | 36
  Linezolid: Cure | 18
  Linezolid: Death: number analyzed (Participants) | 36
  Linezolid: Death | 8
  Tedizolid: Perceived clinical failure/disease progression: number analyzed (Participants) | 4
  Tedizolid: Perceived clinical failure/disease progression | 1
  Tedizolid: Cure: number analyzed (Participants) | 4
  Tedizolid: Cure | 3
  Teicoplanin: Secondary infection requiring regimen change: number analyzed (Participants) | 17
  Teicoplanin: Secondary infection requiring regimen change | 1
  Teicoplanin: De-escalation: number analyzed (Participants) | 17
  Teicoplanin: De-escalation | 2
  Teicoplanin: Cure: number analyzed (Participants) | 17
  Teicoplanin: Cure | 7
  Teicoplanin: Death: number analyzed (Participants) | 17
  Teicoplanin: Death | 2
  Teicoplanin: Other: number analyzed (Participants) | 17
  Teicoplanin: Other | 6
  Telavancin: Cure: number analyzed (Participants) | 1
  Telavancin: Cure | 1
  Vancomycin: AE: number analyzed (Participants) | 65
  Vancomycin: AE | 3
  Vancomycin: Perceived clinical failure/disease progression: number analyzed (Participants) | 65
  Vancomycin: Perceived clinical failure/disease progression | 1
  Vancomycin: Isolation of a resistant pathogen: number analyzed (Participants) | 65
  Vancomycin: Isolation of a resistant pathogen | 5
  Vancomycin: Preference for empiric coverage: number analyzed (Participants) | 65
  Vancomycin: Preference for empiric coverage | 6
  Vancomycin: Secondary infection requiring regimen change: number analyzed (Participants) | 65
  Vancomycin: Secondary infection requiring regimen change | 1
  Vancomycin: Switch to oral therapy: number analyzed (Participants) | 65
  Vancomycin: Switch to oral therapy | 1
  Vancomycin: De-escalation: number analyzed (Participants) | 65
  Vancomycin: De-escalation | 10
  Vancomycin: Cure: number analyzed (Participants) | 65
  Vancomycin: Cure | 30
  Vancomycin: Death: number analyzed (Participants) | 65
  Vancomycin: Death | 2
  Vancomycin: Other: number analyzed (Participants) | 65
  Vancomycin: Other | 8
  Rifaximin: Cure: number analyzed (Participants) | 1
  Rifaximin: Cure | 1
  Metronidazole: Perceived clinical failure/disease progression: number analyzed (Participants) | 59
  Metronidazole: Perceived clinical failure/disease progression | 1
  Metronidazole: Preference for empiric coverage: number analyzed (Participants) | 59
  Metronidazole: Preference for empiric coverage | 4
  Metronidazole: De-escalation: number analyzed (Participants) | 59
  Metronidazole: De-escalation | 8
  Metronidazole: Cure: number analyzed (Participants) | 59
  Metronidazole: Cure | 32
  Metronidazole: Death: number analyzed (Participants) | 59
  Metronidazole: Death | 7
  Metronidazole: Other: number analyzed (Participants) | 59
  Metronidazole: Other | 11
  Ofloxacin ear drops: Cure: number analyzed (Participants) | 1
  Ofloxacin ear drops: Cure | 1
  Clofazimine: Other: number analyzed (Participants) | 1
  Clofazimine: Other | 1
  Ethambutol: Other: number analyzed (Participants) | 1
  Ethambutol: Other | 1
  Isoniazid: Other: number analyzed (Participants) | 2
  Isoniazid: Other | 2

14. Primary Outcome: Number of Participants Whose Samples Were Taken for Clinical Microbiological Evaluation After End of Ceftazidime-Avibactam Therapy: Microbiology Outcomes Dataset (MOD) Population
Description: The number of participants whose samples were taken for clinical microbiological evaluation after end of ceftazidime-avibactam therapy were reported in this outcome measure.
Time Frame: From end of index therapy up to 60 days after hospital discharge, in-hospital death, withdrawal from study, or lost to follow-up, whichever occurred first maximum of 464 days (from the data evaluated in approximately 40 months of the study)
Population: MOD population included all participants with at least 72 hours exposure to ceftazidime-avibactam, identification of one or more pathogens before the start of ceftazidime-avibactam treatment, and at least one non-missing microbiological outcome. Not all participants of MOD population had data collected after end of ceftazidime-avibactam therapy. Hence, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 20
Participants | 20

15. Primary Outcome: Number of Participants Classified According to Type of Specimen Taken for Clinical Microbiological Evaluation After End of Ceftazidime-Avibactam Therapy: MOD Population
Description: The number of participants classified according to the type of specimen taken for clinical microbiological evaluation after end of ceftazidime-avibactam therapy were reported in this outcome measure. More than 1 type of specimen could have been taken from 1 participant.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 20
Participants
  Blood | 10
  Urine | 4
  Bronchoalveolar lavage | 4
  Sputum | 5
  Abscess drainage | 1
  Swab | 3
  Surgical/biopsy specimen | 1
  Other | 5

16. Primary Outcome: Number of Participants Classified According to the Pathogens Identified From the Microbiological Culture After Treatment Initiation: MOD Population
Description: The number of participants classified according to the pathogens identified from the microbiological culture after treatment initiation were reported in this outcome measure.
Time Frame: After treatment initiation up to 60 days post hospital discharge, in-hospital death, withdrawal from the study, or lost to follow-up, whichever occurred first maximum of 464 days (from the data evaluated in approximately 40 months of the study)
Population: MOD population included all participants with at least 72 hours exposure to ceftazidime-avibactam, identification of one or more pathogens before the start of ceftazidime-avibactam treatment, and at least one non-missing microbiological outcome. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 69
Participants
  Gram-negative: Escherichia coli | 4
  Gram-negative: Klebsiella pneumoniae | 15
  Gram-negative: Proteus mirabilis | 1
  Gram-negative: Acinetobacter baumannii | 6
  Gram-negative: Enterobacter cloacae | 2
  Gram-negative: Enterobacter species (spp) | 1
  Gram-negative: Serratia spp | 2
  Gram-negative: Morganella morganii | 1
  Gram-negative: Pseudomonas aeruginosa | 8
  Gram-negative: Pseudomonas spp | 2
  Gram-negative: Other | 8
  Gram-positive: Staphylococcus spp | 6
  Gram-positive: Enterococcus spp | 14
  Gram-positive: Other | 3
  Anaerobes: Clostridium spp | 1
  Other Bacterial Agent | 1

17. Primary Outcome: Number of Gram-Negative Pathogens According to the Susceptibility to Antibiotics After Treatment Initiation: FAS72+ Population
Description: The number of gram-negative pathogens according to the susceptibility to specific antibiotics after treatment initiation were reported in this outcome measure.
Time Frame: as for outcome 16
Population: as for outcome 9
Measure: Number; unit: Pathogens
Units Other Than Participants: Pathogens
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 24
Number analyzed (Pathogens) | 52
Pathogens
  Aminoglycosides | 39
  Amphenicol | 2
  Carbapenems | 39
  Carbapenems: Doripenem: number analyzed (Pathogens) | 39
  Carbapenems: Doripenem | 13
  Carbapenems: Ertapenem: number analyzed (Pathogens) | 39
  Carbapenems: Ertapenem | 17
  Carbapenems: Imipenem: number analyzed (Pathogens) | 39
  Carbapenems: Imipenem | 31
  Carbapenems: Meropenem: number analyzed (Pathogens) | 39
  Carbapenems: Meropenem | 36
  Cephalosporins | 35
  Cephalosporins: Cefalexin: number analyzed (Pathogens) | 35
  Cephalosporins: Cefalexin | 0
  Cephalosporins: Cefazolin: number analyzed (Pathogens) | 35
  Cephalosporins: Cefazolin | 0
  Cephalosporins: Cefepime: number analyzed (Pathogens) | 35
  Cephalosporins: Cefepime | 12
  Cephalosporins: Cefixime: number analyzed (Pathogens) | 35
  Cephalosporins: Cefixime | 1
  Cephalosporins: Cefotaxime: number analyzed (Pathogens) | 35
  Cephalosporins: Cefotaxime | 13
  Cephalosporins: Cefoxitin: number analyzed (Pathogens) | 35
  Cephalosporins: Cefoxitin | 1
  Cephalosporins: Cefpodoxime: number analyzed (Pathogens) | 35
  Cephalosporins: Cefpodoxime | 0
  Cephalosporins: Ceftaroline: number analyzed (Pathogens) | 35
  Cephalosporins: Ceftaroline | 0
  Cephalosporins: Ceftazidime: number analyzed (Pathogens) | 35
  Cephalosporins: Ceftazidime | 27
  Cephalosporins: Ceftriaxone: number analyzed (Pathogens) | 35
  Cephalosporins: Ceftriaxone | 7
  Cephalosporins: Cefuroxime: number analyzed (Pathogens) | 35
  Cephalosporins: Cefuroxime | 2
  Cephalosporin/beta-lactamase inhibitor | 6
  Cephalosporin/beta-lactamase inhibitor: Ceftazidime/avibactam: number analyzed (Pathogens) | 6
  Cephalosporin/beta-lactamase inhibitor: Ceftazidime/avibactam | 5
  Cephalosporin/beta-lactamase inhibitor: Cefoperazone/sulbactam: number analyzed (Pathogens) | 6
  Cephalosporin/beta-lactamase inhibitor: Cefoperazone/sulbactam | 0
  Cephalosporin/beta-lactamase inhibitor: Ceftolozane/tazobactam: number analyzed (Pathogens) | 6
  Cephalosporin/beta-lactamase inhibitor: Ceftolozane/tazobactam | 1
  Glycopeptides | 0
  Glycylcycline | 4
  Lipopeptides | 0
  Macrolides | 0
  Monobactam | 9
  Nitroimidazole | 0
  Oxazolidinones | 0
  Penicillins | 2
  Penicillins and beta-lactamase inhibitors | 30
  Penicillins and beta-lactamase inhibitors: Ampicillin-sulbactam: number analyzed (Pathogens) | 30
  Penicillins and beta-lactamase inhibitors: Ampicillin-sulbactam | 3
  Penicillins and beta-lactamase inhibitors: Amoxicillin-clavulanate: number analyzed (Pathogens) | 30
  Penicillins and beta-lactamase inhibitors: Amoxicillin-clavulanate | 15
  Penicillins and beta-lactamase inhibitors: Piperacillin-tazobactam: number analyzed (Pathogens) | 30
  Penicillins and beta-lactamase inhibitors: Piperacillin-tazobactam | 14
  Penicillins and beta-lactamase inhibitors: Ticarcillin-clavulanate: number analyzed (Pathogens) | 30
  Penicillins and beta-lactamase inhibitors: Ticarcillin-clavulanate | 3
  Fluoroquinolones | 40
  Streptogramins | 0
  Tetracycline | 0
  Other Agents | 13
  Other Agents: Colistin: number analyzed (Pathogens) | 13
  Other Agents: Colistin | 7
  Other Agents: Trimethoprim: number analyzed (Pathogens) | 13
  Other Agents: Trimethoprim | 0
  Other Agents: Trimethoprim-sulfamethoxazole: number analyzed (Pathogens) | 13
  Other Agents: Trimethoprim-sulfamethoxazole | 6
  Other Agents: Fosfomycin: number analyzed (Pathogens) | 13
  Other Agents: Fosfomycin | 1
  Other Agents: Nitrofurantoin: number analyzed (Pathogens) | 13
  Other Agents: Nitrofurantoin | 0

18. Primary Outcome: Number of Gram-Negative Pathogens According to the Multi-Drug Resistance After Treatment Initiation: FAS72+ Population
Description: Multi-drug resistance was defined as the isolate being non-susceptible to at least one agent in more than or equal to (>=) 3 antimicrobial categories, excluding the therapeutic classes to which the pathogen was intrinsically resistant. The number of gram-negative pathogens classified according to the antibiotic resistance to specified antibiotics after treatment initiation were reported in this outcome measure.
Time Frame: as for outcome 16
Population: as for outcome 9
Measure: Number; unit: Pathogens
Units Other Than Participants: Pathogens
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 24
Number analyzed (Pathogens) | 26
Pathogens
  Aminoglycosides | 21
  Amphenicol | 2
  Carbapenems | 25
  Carbapenems: Doripenem: number analyzed (Pathogens) | 25
  Carbapenems: Doripenem | 13
  Carbapenems: Ertapenem: number analyzed (Pathogens) | 25
  Carbapenems: Ertapenem | 12
  Carbapenems: Imipenem: number analyzed (Pathogens) | 25
  Carbapenems: Imipenem | 20
  Carbapenems: Meropenem: number analyzed (Pathogens) | 25
  Carbapenems: Meropenem | 25
  Cephalosporins | 24
  Cephalosporins: Cefalexin: number analyzed (Pathogens) | 24
  Cephalosporins: Cefalexin | 0
  Cephalosporins: Cefazolin: number analyzed (Pathogens) | 24
  Cephalosporins: Cefazolin | 0
  Cephalosporins: Cefepime: number analyzed (Pathogens) | 24
  Cephalosporins: Cefepime | 6
  Cephalosporins: Cefixime: number analyzed (Pathogens) | 24
  Cephalosporins: Cefixime | 1
  Cephalosporins: Cefotaxime: number analyzed (Pathogens) | 24
  Cephalosporins: Cefotaxime | 9
  Cephalosporins: Cefoxitin: number analyzed (Pathogens) | 24
  Cephalosporins: Cefoxitin | 1
  Cephalosporins: Cefpodoxime: number analyzed (Pathogens) | 24
  Cephalosporins: Cefpodoxime | 0
  Cephalosporins: Ceftaroline: number analyzed (Pathogens) | 24
  Cephalosporins: Ceftaroline | 0
  Cephalosporins: Ceftazidime: number analyzed (Pathogens) | 24
  Cephalosporins: Ceftazidime | 24
  Cephalosporins: Ceftriaxone: number analyzed (Pathogens) | 24
  Cephalosporins: Ceftriaxone | 6
  Cephalosporins: Cefuroxime: number analyzed (Pathogens) | 24
  Cephalosporins: Cefuroxime | 1
  Cephalosporin/beta-lactamase inhibitor | 4
  Cephalosporin/beta-lactamase inhibitor: Ceftazidime/avibactam: number analyzed (Pathogens) | 4
  Cephalosporin/beta-lactamase inhibitor: Ceftazidime/avibactam | 4
  Cephalosporin/beta-lactamase inhibitor: Cefoperazone/sulbactam: number analyzed (Pathogens) | 4
  Cephalosporin/beta-lactamase inhibitor: Cefoperazone/sulbactam | 0
  Cephalosporin/beta-lactamase inhibitor: Ceftolozane/tazobactam: number analyzed (Pathogens) | 4
  Cephalosporin/beta-lactamase inhibitor: Ceftolozane/tazobactam | 0
  Cephalosporin/beta-lactamase inhibitor: Glycopeptides: number analyzed (Pathogens) | 4
  Cephalosporin/beta-lactamase inhibitor: Glycopeptides | 0
  Glycylcycline | 2
  Lipopeptides | 0
  Macrolides | 0
  Monobactam | 9
  Nitroimidazole | 0
  Oxazolidinones | 0
  Penicillins | 1
  Penicillins and beta-lactamase inhibitors | 21
  Penicillins and beta-lactamase inhibitors: Ampicillin-sulbactam: number analyzed (Pathogens) | 21
  Penicillins and beta-lactamase inhibitors: Ampicillin-sulbactam | 1
  Penicillins and beta-lactamase inhibitors: Amoxicillin-clavulanate: number analyzed (Pathogens) | 21
  Penicillins and beta-lactamase inhibitors: Amoxicillin-clavulanate | 12
  Penicillins and beta-lactamase inhibitors: Piperacillin-tazobactam: number analyzed (Pathogens) | 21
  Penicillins and beta-lactamase inhibitors: Piperacillin-tazobactam | 8
  Penicillins and beta-lactamase inhibitors: Ticarcillin-clavulanate: number analyzed (Pathogens) | 21
  Penicillins and beta-lactamase inhibitors: Ticarcillin-clavulanate | 3
  Fluoroquinolones | 24
  Streptogramins | 0
  Tetracycline | 0
  Other Agents | 5
  Other Agents: Colistin: number analyzed (Pathogens) | 5
  Other Agents: Colistin | 4
  Other Agents: Trimethoprim: number analyzed (Pathogens) | 5
  Other Agents: Trimethoprim | 0
  Other Agents: Trimethoprim-sulfamethoxazole: number analyzed (Pathogens) | 5
  Other Agents: Trimethoprim-sulfamethoxazole | 1
  Other Agents: Fosfomycin: number analyzed (Pathogens) | 5
  Other Agents: Fosfomycin | 0
  Other Agents: Nitrofurantoin: number analyzed (Pathogens) | 5
  Other Agents: Nitrofurantoin | 0

19. Primary Outcome: Number of Participants Classified According to Type of Clinical Evaluation Outcome at Initial Hospitalization: Clinical Outcomes Dataset (COD) Population
Description: The number of participants classified according to type of clinical evaluation outcome as success, failure or indeterminate. Success: resolution of all signs and symptoms of infection with no need for escalation of antimicrobials for gram-negative coverage. Failure: inadequate response to ceftazidime-avibactam therapy or resistant, worsening, or new recurrent signs and symptoms at the end of ceftazidime-avibactam therapy. Indeterminate: there was not enough information to conclude whether the antibiotic regimen containing ceftazidime-avibactam was a clinical failure or a success.
Time Frame: At initial hospitalization (from the data evaluated in approximately 40 months of this study)
Population: COD population included all participants with at least 72 hours exposure to ceftazidime-avibactam and at least one non-missing clinical outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants
  Success | 399
  Failure | 60
  Indeterminate | 57

20. Primary Outcome: Number of Participants Classified According to Type of Clinical Evaluation Outcome 60 Days Post-Discharge: Clinical Outcomes Dataset (COD) Population
Description: as for outcome 19
Time Frame: 60 days after hospital discharge (from the data evaluated in approximately 40 months of this study)
Population: COD population included all participants with at least 72 hours exposure to ceftazidime-avibactam and at least one non-missing clinical outcome. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 317
Participants
  Success | 266
  Failure | 27
  Indeterminate | 24

21. Primary Outcome: Number of Participants Classified According to Type of Clinical Evaluation Outcome 60 Days Post-Treatment: Clinical Outcomes Dataset (COD) Population
Description: as for outcome 19
Time Frame: 60 days post treatment (from the data evaluated in approximately 40 months of this study)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 374
Participants
  Success | 311
  Failure | 32
  Indeterminate | 31

22. Primary Outcome: Number of Participants With Microbiological Treatment Outcome as Success: MOD Population
Description: The number of participants with microbiological treatment outcome as success were reported in this outcome measure. Success was defined as: absence of causative pathogen from appropriately obtained specimens at the site of infection.
Time Frame: Up to 14 days post first dose of ceftazidime-avibactam (from the data evaluated in approximately 40 months of the study)
Population: Planned analysis of this outcome measure was cancelled on approval of Scientific Steering Committee as few participants had microbiological cultures after the start of ceftazidime-avibactam.
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 0

23. Primary Outcome: Number of Participants Classified According to Antibiotics Used for Current Infection Before Ceftazidime-Avibactam: FAS72+ Population
Description: The number of participants classified according to antibiotics used (Yes or No) for current infection before ceftazidime-avibactam were reported in this outcome measure.
Time Frame: Up to 90 days prior to index date (from the data evaluated in approximately 40 months of this study)
Population: FAS72+ population included all participants with at least 72 hours of exposure to ceftazidime-avibactam.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants
  Yes | 397
  No | 119

24. Primary Outcome: Number of Participants Classified According to Reason for Discontinuation for Prior Antibiotic Therapy: FAS72+ Population
Description: The number of participants classified according to reason for discontinuing for prior antibiotic therapy were reported in this outcome measure. One participant could have more than 1 reason of discontinuation for prior antibiotic therapy.
Time Frame: Up to 90 days prior to index date (from the data evaluated in approximately 40 months of this study)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 389
Participants
  AE | 11
  Perceived clinical failure/disease progression | 134
  Isolation of a resistant pathogen | 236
  Preference for empiric coverage | 32
  Secondary infection requiring regimen change | 35
  Switch to oral therapy | 4
  De-escalation | 58
  Cure | 53
  Death | 11
  Other | 69

25. Primary Outcome: Percentage of Participants Who Died During Index Hospitalization
Description: In hospital-mortality was defined as deaths occurring after treatment initiation but before hospital discharge. The percentage of participants who died during index hospitalization were reported in this outcome measure.
Time Frame: During index hospitalization, maximum of 418 days (from the data evaluated in approximately 40 months of this study)
Population: FAS72+ population included all participants with at least 72 hours of exposure to Ceftazidime-avibactam.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Percentage of participants | 23.1 [19.5 to 26.9]

26. Primary Outcome: Percentage of Participants Who Died Within the 30 Days After Hospital Discharge (Including In-Hospital Mortality): FAS72+ Population
Description: 30-day mortality was defined as deaths occurred from index treatment up to within 30 days after hospital discharge including in-hospital mortality.
Time Frame: From index treatment up to 30 days post hospital discharge, maximum of 434 days (from the data evaluated in approximately 40 months of this study)
Population: FAS72+ population included all participants with at least 72 hours of exposure to Ceftazidime-avibactam.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Percentage of participants | 24.6 [21.0 to 28.6]

27. Primary Outcome: Percentage of Participants Who Died Within 60 Days After Hospital Discharge (Including In-Hospital Mortality): FAS72+ Population
Description: 60-day mortality was defined as deaths occurred from index treatment up to within 60 days after hospital discharge including in-hospital mortality.
Time Frame: From index treatment up to 60 days post hospital discharge, maximum of 434 days (from the data evaluated in approximately 40 months of this study)
Population: FAS72+ population included all participants with at least 72 hours of exposure to Ceftazidime-avibactam.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Percentage of participants | 27.9 [24.1 to 32]

28. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. AE included both SAEs and non-SAEs. SAE was defined as any untoward medical occurrence at any dose that: resulted in death, was life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required hospitalization or prolongation of existing hospitalization. Only AEs and SAEs with explicit attribution to ceftazidime-avibactam that appeared in the reviewed information and scenarios involving drug exposure to ceftazidime-avibactam, which included exposure during pregnancy, exposure during breastfeeding, medication error, overdose, misuse, extravasation, lack of efficacy and occupational exposure associated with the use of ceftazidime-avibactam were collected in the study.
Time Frame: From index date up to 60 days after hospital discharge, in-hospital death, withdrawal from the study, or lost to follow-up, whichever occurred first maximum of 464 days (from the data evaluated in approximately 40 months of the study)
Population: FAS population included all enrolled participants meeting the study eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 569
Participants
  Any adverse event | 6
  Any serious adverse event | 5

29. Primary Outcome: Duration of Hospital Stay: FAS72+ Population
Description: Hospital length of stay (LOS) was defined as date of hospital discharge minus date of hospital admission plus 1. The duration of hospital stay of participants were reported in this outcome measure.
Time Frame: From index date up to hospital discharge, in-hospital death, withdrawal from the study, or lost to follow-up, whichever occurred first maximum of 418 days (from the data evaluated in approximately 40 months of the study)
Population: as for outcome 9
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 514
Days | 36.0 [3 to 418]

30. Primary Outcome: Total Duration of ICU Stay: FAS72+ Population
Description: Duration of ICU stay was defined as date of ICU discharge minus date of ICU admission plus 1. The total duration of ICU stay of participants were reported in this outcome measure.
Time Frame: During index hospitalization, maximum up to 418 days (from the data evaluated in approximately 40 months of the study)
Population: as for outcome 9
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 275
Days | 24.0 [1 to 405]

31. Primary Outcome: Number of Participants Readmitted to the Hospital During the 30 Days After Initial Discharge: FAS72+ Population
Description: The number of participants readmitted to the hospital during the 30 days after initial discharge were reported in this outcome measure.
Time Frame: Up to 30 days after initial discharge (from the data evaluated in approximately 40 months of the study)
Population: FAS72+ population included all participants with at least 72 hours of exposure to Ceftazidime-avibactam.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants | 111

32. Primary Outcome: Number of Participants Readmitted to the Hospital During the 60 Days After Initial Discharge: FAS72+ Population
Description: The number of participants readmitted to the hospital during the 60 days after initial discharge were reported in this outcome measure.
Time Frame: Up to 60 days after initial discharge (from the data evaluated in approximately 40 months of the study)
Population: FAS72+ population included all participants with at least 72 hours of exposure to Ceftazidime-avibactam.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants | 53

33. Primary Outcome: Number of Participants Classified According to Reason for Readmission to the Hospital: FAS72+ Population
Description: The number of participants classified according to the reason for readmission to the hospital were reported in this outcome measure. One participant could have more than 1 reason for readmission to the hospital.
Time Frame: At readmission to the hospital, up to maximum of 60 days post initial hospital discharge (from the data evaluated in approximately 40 months of the study)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 137
Participants
  Unrelated to the infection | 98
  Infection recurrence | 25
  Secondary infection | 17
  Unknown | 6

34. Primary Outcome: Number of Participants Classified According to the Healthcare Resource Utilized During the Hospitalization: FAS72+ Population
Description: The number of participants classified according to the healthcare resource utilization during the hospitalization were reported in this outcome measure. One participant could have utilized more than 1 healthcare resource during hospitalization.
Time Frame: During index hospitalization maximum of 418 days (from the data evaluated in approximately 40 months of the study)
Population: FAS72+ population included all participants with at least 72 hours of exposure to Ceftazidime-avibactam.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 516
Participants
  Mechanical ventilation | 161
  Hemodialysis | 80
  CT/MRI imaging | 273
  Tracheostomy | 83
  Surgical intervention | 169
  Percutaneous procedures | 149
  Other | 73

35. Primary Outcome: Number of Participants Classified According to All Wards Attended During Hospitalization: FAS72+ Population
Description: The number of participants classified according to all wards attended during hospitalization were reported in this outcome measure.
Time Frame: During index hospitalization maximum of 418 days (from the data evaluated in approximately 40 months of the study)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-avibactam
Number analyzed (Participants) | 515
Participants
  Surgical | 101
  Medical | 195
  Onco-hematology | 58
  Infectious disease | 27
  ICU | 116
  Other | 18

ADVERSE EVENTS:
Time Frame: From index date up to 60 days after hospital discharge, in-hospital death, withdrawal from the study, or lost to follow-up, whichever occurred first (up to maximum of 464 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Only SAEs and non-SAEs with an explicit attribution to or associated with use of ceftazidime-avibactam from the data captured in medical records were collected in this study.
Arm/Group | Ceftazidime-avibactam
All-Cause Mortality (participants affected / at risk) | 170/569
Serious Adverse Events (participants affected / at risk) | 5/569
Other Adverse Events (participants affected / at risk) | 2/569
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftazidime-avibactam (N=569)
Multiple organ dysfunction syndrome (General disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Altered state of consciousness (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftazidime-avibactam (N=569)
Diarrhoea (Gastrointestinal disorders) | 1
Blurred vision (Eye disorders) | 1
Confusional state (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03923426/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT03923426/SAP_001.pdf